CLINICAL TRIAL: NCT03493334
Title: Impacto do Feedback Visual da região Posterior da Coluna Cervical, na Intensidade da Dor e Amplitude de Movimento, em Utentes Com Dor Cervical crónica idiopática
Brief Title: Visual Feedback in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-CED/2018
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual feedback (Experimental): Participants in this group will receive visual feedback of their neck when performing 10 repetitions of each of neck movements (flexion, extension, side-flexion and rotation).
  Interventions: Other: Visual feedback
- No visual feedback (Active Comparator): Participants in this group will perform 10 repetitions of each of neck movements (flexion, extension, side-flexion and rotation) without feedback.
  Interventions: Other: No visual feedback

INTERVENTIONS:
Other: Visual feedback — Visual feedback of the neck will be given to participants using two mirrors while performing neck movements.
  Arms: Visual feedback
Other: No visual feedback — Participants will be asked to perform active movements of their neck with the mirrors covered.
  Arms: No visual feedback

SUMMARY:
The objective of this study is to evaluate the impact of visual feedback of the posterior region of the cervical spine on pain intensity and range of motion.

DETAILED DESCRIPTION:
60 patients with chronic idiopathic neck pain will be randomly assigned into one of two groups: a group receiving visual feedback when performing 10 repetitions of each of neck movements (flexion, extension, side-flexion and rotation) and a group performing the same task without visual feedback. Participants will be assessed for pain intensity, pain location, disability, range of motion, kinesiophobia, catastrophizing and anxiety both at baseline and after visual the intervention (i.e., neck movements with and without visual feedback).

ELIGIBILITY:
Inclusion Criteria:

* To have idiopathic neck pain defined as neck pain unrelated to any known pathology or lesion felt at least once a week in the last 3 months, located between the nuchal line and a horizontal line passing through T1 and pain intensity of at least 3 in the visual analogue scale.

Exclusion Criteria:

* History of cervical or facial trauma, radiculopathy, history of surgery in the vertebral segment in question, congenital anomalies involving the spine (cervical, thoracic and lumbar spine) or any neurological or rheumatic pathology, and, finally, evidence of significant visual changes, or of deficits not corrected by lenses or glasses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity | Baseline
  Measured using a 10 cm visual analogue scale
Neck pain intensity | Immediately after the intervention (at 30 minutes)
  Measured using a 10 cm visual analogue scale

SECONDARY OUTCOMES:
Pain location | Baseline
  Measured using a body chart
Pain location | Immediately after the intervention (at 30 minutes)
  Measured using a body chart
Time for pain to return to baseline levels | Immediately after the intervention (at 30 minutes)
  Measured with a chronometer
Pain disability | Baseline
  Measured using the Neck Disability Questionnaire (range: 0-50 and higher scores are indicative of more disability)
Pain disability | Immediately after the intervention (at 30 minutes)
  Measured using the Neck Disability Questionnaire (range: 0-50 and higher scores are indicative of more disability)
Neck range of motion | Baseline
  Measured using a goniometer
Neck range of motion | Immediately after the intervention (at 30 minutes)
  Measured using a goniometer
Kinesiophobia | Baseline
  Measured using the Tampa Scale of Kinsesiophobia (Range: 13-52 and higher values are indicative of a higher fear of movement.
Kinesiophobia | Immediately after the intervention (at 30 minutes)
  Measured using the Tampa Scale of Kinsesiophobia (Range: 13-52 and higher values are indicative of a higher fear of movement.
Catastrophyzing | Baseline
  Measured using the Pain Catastrophyzing Scale (range: 0-52 and higher scores and indicative of higher pain catastrophyzing)
Catastrophyzing | Immediately after the intervention (at 30 minutes)
  Measured using the Pain Catastrophyzing Scale (range: 0-52 and higher scores and indicative of higher pain catastrophyzing)
Anxiety | Baseline
  Measured using the State-Trait Anxiety Scale, which consists of 2 sub-scales, one measures trait anxiety and the other measures state anxiety; both scales have an independent score that ranges from 20 to 80 and higher scores are indicative of higher anxiety.
Anxiety | Immediately after the intervention (at 30 minutes)
  Measured using the State-Trait Anxiety Scale, which consists of 2 sub-scales, one measures trait anxiety and the other measures state anxiety; both scales have an independent score that ranges from 20 to 80 and higher scores are indicative of higher anxiety.
Neck perception | Baseline
  Assessed by asking participants to draw their neck as they perceive it to be
Neck perception | Immediately after the intervention (at 30 minutes)
  Assessed by asking participants to draw their neck as they perceive it to be

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Principal Investigator — Aveiro University
Locations (1):
- Clínica de Diagnóstico e Terapêutica - Hellman, Lda, Figueira da Foz Municipality, Portugal

IPD SHARING:
Plan to Share IPD: No